CLINICAL TRIAL: NCT06669910
Title: Investıgatıon of Temporomandıbular Dysfunctıon in Patıents Wıth Breast Cancer-Related Lymphedema
Status: Completed | Type: Observational
Sponsor: arife akbulut (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, arife akbulut, LECTURER, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Other Study IDs: AYBU-AKBULUT-001
Record Dates: First submitted 2024-08-14; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- mild TMD
  Interventions: Other: only assesment
- moderate TMD
  Interventions: Other: only assesment
- advanced TMD
  Interventions: Other: only assesment

INTERVENTIONS:
Other: only assesment — only assesment

SUMMARY:
This study is the first study to examine temporomandibular joint dysfunction (TMD) in patients with breast cancer. The aim of the study was to investigate the relationship between lymphedema (LÖ) and TMD in patients with breast cancer. Socio-demographic characteristics of 38 individuals included in the study were recorded. Patients were divided into stage 0, 1 and 2 groups according to their LÖ stage and mild, moderate and advanced groups according to their TMD levels. In the evaluation of severity of lymphedema, Symptoms and Signs of TMD, pain threshold and tolerance assessment and normal range of motion, anxiety and depression, posture analysis environmental measurement, Craniomandibular Dysfunction Index for Clinical, Visual Analogue Scale (VAS) and algometer , goniometer and inclinometer, Turkish version of the Hospital Anxiety and Depression Scale (HAD) ,photogrammetric assessment method and inclinometer were used

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-75 years who were treated for unilateral breast cancer and developed breast cancer-related LE were included in the study

Exclusion Criteria:

* Patients with general joint diseases affecting the head and neck region that may cause TMD (e.g. rheumatoid arthritis),
* jaw fracture,
* trauma or orthognathic surgery history,
* cervical disc herniation,
* congenital disease,
* facial paralysis,
* patients who have been treated for TMD for the last 3 months and patients who use antidepressant drugs were excluded.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients who were treated for unilateral breast cancer and developed breast cancer-related LE
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
temporomandibular dysfunction | through study completion, an average of 1 year
  The Clinical Craniomandibular Dysfunction Index (CDI) was used. CDI consists of five components including limited mandibular normal joint motion (RMJ), pain during mandibular RMJ, pain during TMJ palpation, pain during palpation of masticatory muscles and pain during mandibular function. 3 points can be given for each component as 0, 1 or 5 points and individuals are graded as no TMD (0 points), mild TMD (1-4 points), moderate TMD (5-9 points) and severe TMD (10-25 points) according to the scores received.
lymhedema | through study completion, an average of 1 year
  It was determined according to the criteria determined by the International Lymphology Association . To determine the severity of LE, circumference measurements were taken from both arms at 4 cm intervals. If the difference between the two extremities was up to 1.5 cm, it was classified as "normal", between 1.5-3 cm as "mild", between 3-5 cm as "moderate" and over 5 cm as "severe" LE

SECONDARY OUTCOMES:
pain | through study completion, an average of 1 year
  The pain was assessed with the Visual Analog Scale (VAS) at rest and activity. Patients were asked to mark the point that best described their pain on a 10 cm line (0: no pain, 10: unbearable pain). The pain intensity with activity was assessed during mouth opening, mouth closing and 60 seconds of gum chewing. Patients were asked to chew gum using both sides for 60 seconds. At the end of this period, patients evaluated their pain in the TMJ according to the VAS
posture | through study completion, an average of 1 year
  Kyphosis and lordosis angles of the patients were measured with Baseline® Digital inclinometer while the patients were standing in a comfortable position. "Posture Analysis Method with Photography" was used.
Measurement of range of motion of cervical joints and shoulder joint | through study completion, an average of 1 year
  The measurements were made with a Baseline® universal goniometer with a plastic 360 degree quadrant. Flexion, extension, right-left lateral flexion and rotation angles for the cervical region, and flexion, abduction, external and internal rotation ROM angles for the shoulder joint were measured. The measurements were made in the sitting position for the cervical region and in the supine position for the shoulder. Each measurement was repeated 3 times and the average values were recorded.
anxiety-depression | through study completion, an average of 1 year
  The Turkish version of the Hospital Anxiety and Depression Scale (HAD) was used. HAD is a 4-point Likert-type scale with a score between 0 and 21, consisting of 14 questions, 7 of which evaluate anxiety and 7 of which evaluate depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Arife Akbulut, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akbulut Bayrak A, Tekbudak MY, Gultekin S, Keser I. Investigation of temporomandibular dysfunction in patients with breast cancer-related lymphedema. Support Care Cancer. 2025 May 7;33(6):455. doi: 10.1007/s00520-025-09500-y. PMID 40332621